CLINICAL TRIAL: NCT04947800
Title: Exploring the Dose-Response Effect of Adjunctive Acupuncture on Pulmonary Rehabilitation: A Pilot Study
Brief Title: Acupuncture to Enhance for Pulmonary Rehab
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1) Closure of pulm rehab program from which patients were recruited 2) recurrent IRB delays
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Academy of Medical Acupuncture (Unknown)
Responsible Party: Principal Investigator, James E. Stahl, Principal Investigator; Staff Physician, General Internal Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY02000887
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told which weeks they are receiving the active acupuncture versus the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm A: 12 week intervention, 8 week control (Experimental): Electro acupuncture (EA) intervention will be administered for 12 weeks to the Lung Mu-Shu points and St36 which are related to lung function and general function. The EA control intervention will be administered for 8 weeks and will use Lv7 and Gb 26 which are near the other points but not traditionally related to lung function or general function.
  Interventions: Device: Pulmonary rehabilitation program + EA Lung Mu-Shu+ St36; Device: Pulmonary rehabilitation program + Lv7/Gb26
- Arm B: 8 week intervention, 12 week control (Experimental): Electro acupuncture (EA) intervention will be administered for 8 weeks to the Lung Mu-Shu points and St36 which are related to lung function and general function. The EA control intervention will be administered for 12 weeks and will use Lv7 and Gb 26 which are near the other points but not traditionally related to lung function or general function.
  Interventions: Device: Pulmonary rehabilitation program + EA Lung Mu-Shu+ St36; Device: Pulmonary rehabilitation program + Lv7/Gb26
- Arm C: 4 week intervention, 16 week control (Experimental): Electro acupuncture (EA) intervention will be administered for 4 weeks to the Lung Mu-Shu points and St36 which are related to lung function and general function. The EA control intervention will be administered for 16 weeks and will use Lv7 and Gb 26 which are near the other points but not traditionally related to lung function or general function.
  Interventions: Device: Pulmonary rehabilitation program + EA Lung Mu-Shu+ St36; Device: Pulmonary rehabilitation program + Lv7/Gb26

INTERVENTIONS:
Device: Pulmonary rehabilitation program + EA Lung Mu-Shu+ St36 — Standard of care pulmonary rehabilitation program plus electro-acupuncture with mA electricity at varying frequencies to the Lung Mu-Shu points and St36 points
Device: Pulmonary rehabilitation program + Lv7/Gb26 — Standard of care pulmonary rehabilitation program plus electro-acupuncture with mA electricity at varying frequencies to the Lv7/Gb26 points

SUMMARY:
The investigator is investigating if acupuncture may improve pulmonary function, exercise tolerance, stress and modulate the inflammatory effects of chronic obstructive pulmonary disease (COPD). The investigator would like to measure the effect of the combination of acupuncture with standard pulmonary rehab in patients with COPD.

DETAILED DESCRIPTION:
Participation in this study may last 3 months. The experimental intervention is electro-acupuncture. Electro-acupuncture is similar to Transcutaneous Electrical Nerve Stimulation (TENS) where a very small current of electricity is applied, in this case to specific acupuncture points. The intervention will be applied by a trained physician-acupuncturist. The treatment itself would be applied for 20 minutes prior to regularly scheduled pulmonary rehab session. All participants will receive electro-acupuncture for the duration of the study. Because the investigators are interested in the effect of dose, participants will be randomized to 4, 8 or 12 weeks of "active pulmonary" acupuncture versus "control" acupuncture. One third of the participants will be asked to undergo the intervention for 4 weeks, one third will be asked to undergo the intervention for 8 weeks and one third will be asked to undergo the intervention for 12 weeks. Intervention acupuncture needles will be placed on what are thought to be active points for helping lung function, control acupuncture needles will be placed in neutral locations. Participants will not be told which weeks they are receiving the active acupuncture versus the control. Information relating to pulmonary and physical function, standard blood markers of inflammation, and survey responses at the beginning, during and after the intervention will be collected. During the experimental period participants will be asked to fill out surveys on quality of life, pulmonary function and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Qualify to participate in the pulmonary rehab program at DHMC

Exclusion Criteria:

* Severe cognitive impairment
* Active pulmonary exacerbation
* Unstable cardiopulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Stahl, MD, CM, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Started | 8 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — 1) Closure of pulm rehab program from which patients were recruited 2) recurrent IRB delays | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1) Closure of pulm rehab program from which patients were recruited 2) recurrent IRB delays
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control | Total
Number analyzed (Participants) | 8 | 0 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 5 |  |  | 5
Age, Continuous [Mean (Full Range); unit: years] | 67.9 [46 to 84] |  |  | 67.9 [46 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 |  |  | 5
  Male | 3 |  |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 0 |  |  | 0
  White | 8 |  |  | 8
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 |  |  | 8
Pulmonary Function Test (FEV1) [Mean (Full Range); unit: Liters] | 1.38 [.96 to 1.95] |  |  | 1.38 [.96 to 1.96]

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume in One Second (FEV1)
Description: Change in Forced expiratory volume in one second (FEV1) as measures by spirometry test
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: Only baseline data was collected for Arm A. The study was closed before any data was collected for any other timepoints or Arms.
Measure: Mean (Full Range); unit: Liters
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 8 | 0 | 0
Liters | 1.38 [.96 to 1.95] |  |

2. Primary Outcome: Change in Forced Vital Capacity (FVC)
Description: Change in Forced vital capacity (FVC) as measures by spirometry test
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: The study was closed before any data was collected for any outcome measure aside from "Change in Forced expiratory volume in one second (FEV1)"
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change in Number of Eosinophils
Description: Change in number of eosinophils as measured in blood samples
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Change in Number of Neutrophil
Description: Change in number of neutrophil as measured in blood samples
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Change in Number of C Reactive Protein
Description: Change in number of C reactive protein as measured in blood samples
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

6. Primary Outcome: Quality of Life Relating to Dyspnea as Measured by Borg Scales
Description: The Borg Dyspnea Scale scores range from 0 to 10, measuring subjective respiratory exertion with higher scores being worse
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Change in Health Related Quality of Life as Measured by the St. George's Respiratory Questionnaire
Description: The St. George's Respiratory Questionnaire scores range from 0 to 100, with higher scores indicating more limitations. The 50-item questionnaire was developed to measure health status (quality of life) in patients with diseases of airways obstruction.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Change in Health Related Quality of Life as Measure by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire-9 scale questionnaire measures the level of depression. Score range is 0 to 27 points. Higher scores mean more severe depression.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: Change in 6-minute Walk Distance
Description: Change in maximum distance walked in 6 minutes
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: Incidence of Acute Exacerbations (AE)
Description: Throughout the course of the study acute exacerbations will be recorded and tallied.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and 16 weeks
Population: as for outcome 2
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The study was closed before any data was collected related to Adverse Events. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Arm A: 12 week intervention, 8 week control | Arm B: 8 week intervention, 12 week control | Arm C: 4 week intervention, 16 week control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Institutional challenges with IRB and and cutting pulmonary rehab program prevented this trial from being completed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04947800/Prot_SAP_000.pdf